CLINICAL TRIAL: NCT00767923
Title: Clinical Validation of HyperMed OxyVu Tissue Oximeter for Assessing Level of Amputation With Comparison to Other Modalities
Brief Title: Validation of OxyVu for Assessing Level of Amputation With Comparison to Other Modalities
Acronym: LOA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HyperMed (Industry)
Collaborators: Carl T. Hayden VA Medical Center (U.S. Federal Agency)
Responsible Party: Kevin Schomacker, PhD, HyperMed, Inc.
Other Study IDs: 2008-011
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Critical Limb Ischemia
Keywords: hyperspectral imaging; tissue oxygenation; foot amputation; critical limb ischemia; tissue necrosis
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Correlation of(OxyVu) values to to ABI, TBP, and TCOM in patients scheduled for foot level amputation because of critical limb ischemia, infection, or tissue necrosis.

DETAILED DESCRIPTION:
The purpose of this clinical study is to correlate tissue oxygenation values measured with a hyperspectral imaging system (OxyVu) to Ankle Brachial Indices (ABI), toe pressures (TBP), and transcutaneous oxygen monitoring (TCOM) in patients scheduled for foot level amputation because of critical limb ischemia, infection, or tissue necrosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age, males and females, varying skin tones, varying racial origins, and with and without diabetes.
* Patients scheduled for foot level amputation because of critical limb ischemia, infection, or tissue necrosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 to 85 years of age, males and females, varying skin tones, varying racial origins, and with and without diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Assess predictive value for healing by 8 weeks of OxyVu, ABI, TBI and TCOM measured prior to amputation. OxyVu readings for oxyhemoglobin, deoxyhemoglobin and oxygen saturation will be compared to healing potential predicted from ABI, TBI, and TCOM. | 8 weeks

SECONDARY OUTCOMES:
Collect additional interventions required through review of patient medical records at 12 months | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Frykberg, DPM MPH, Principal Investigator — Carl T. Hayden VA Medical Center
Locations (1):
- Carl T Hayden VA Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Second European Consensus Document on chronic critical leg ischemia. Eur J Vasc Surg. 1992 May;6 Suppl A:1-32. No abstract available. PMID 1533191
- [Background] Deerochanawong C, Home PD, Alberti KG. A survey of lower limb amputation in diabetic patients. Diabet Med. 1992 Dec;9(10):942-6. doi: 10.1111/j.1464-5491.1992.tb01736.x. PMID 1478041
- [Background] Frykberg RG. Guidelines for diabetic foot care. Foot Ankle Int. 2000 Jul;21(7):616. doi: 10.1177/107110070002100716. No abstract available. PMID 10919631
- [Background] Ramsey SD, Newton K, Blough D, McCulloch DK, Sandhu N, Reiber GE, Wagner EH. Incidence, outcomes, and cost of foot ulcers in patients with diabetes. Diabetes Care. 1999 Mar;22(3):382-7. doi: 10.2337/diacare.22.3.382. PMID 10097914
- [Background] Harrington C, Zagari MJ, Corea J, Klitenic J. A cost analysis of diabetic lower-extremity ulcers. Diabetes Care. 2000 Sep;23(9):1333-8. doi: 10.2337/diacare.23.9.1333. PMID 10977028
- [Background] Greenman RL, Panasyuk S, Wang X, Lyons TE, Dinh T, Longoria L, Giurini JM, Freeman J, Khaodhiar L, Veves A. Early changes in the skin microcirculation and muscle metabolism of the diabetic foot. Lancet. 2005 Nov 12;366(9498):1711-7. doi: 10.1016/S0140-6736(05)67696-9. PMID 16291064
- [Background] Zuzak KJ, Schaeberle MD, Gladwin MT, Cannon RO 3rd, Levin IW. Noninvasive determination of spatially resolved and time-resolved tissue perfusion in humans during nitric oxide inhibition and inhalation by use of a visible-reflectance hyperspectral imaging technique. Circulation. 2001 Dec 11;104(24):2905-10. doi: 10.1161/hc4901.100525. PMID 11739304
- [Background] Khaodhiar L, Dinh T, Schomacker KT, Panasyuk SV, Freeman JE, Lew R, Vo T, Panasyuk AA, Lima C, Giurini JM, Lyons TE, Veves A. The use of medical hyperspectral technology to evaluate microcirculatory changes in diabetic foot ulcers and to predict clinical outcomes. Diabetes Care. 2007 Apr;30(4):903-10. doi: 10.2337/dc06-2209. Epub 2007 Feb 15. PMID 17303790
- [Background] Benaron DA, Parachikov IH, Friedland S, Soetikno R, Brock-Utne J, van der Starre PJ, Nezhat C, Terris MK, Maxim PG, Carson JJ, Razavi MK, Gladstone HB, Fincher EF, Hsu CP, Clark FL, Cheong WF, Duckworth JL, Stevenson DK. Continuous, noninvasive, and localized microvascular tissue oximetry using visible light spectroscopy. Anesthesiology. 2004 Jun;100(6):1469-75. doi: 10.1097/00000542-200406000-00019. PMID 15166566
- See also: Sponsor and OxyVu technology website — http://www.hypermed-inc.com